CLINICAL TRIAL: NCT00925873
Title: A Randomized Study of Fludarabine in Part of Induction and Postremission Treatment for de Novo Acute Myeloid Leukaemia in Elderly Patients
Brief Title: GOELAMS SA4 Study: the Role of Fludarabine in the Treatment of Acute Myeloid Leukemia in the Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Schering SA (Unknown); Novartis (Industry)
Responsible Party: Dr Francis WITZ, GOELAMS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOELAMS SA4
Record Dates: First submitted 2009-03-31; First posted 2009-06-22 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: Fludarabine; AML; elderly patients
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Control arm without fludarabine
  1. Induction course: Ara-C 100mg/m2 days 1-7, idarubicin 8mg/m2 days 1-5, GM-CSF (molgramostim, Novartis) 5 microg/kg days 1 to neutrophil recovery;
  2. Consolidation course: Ara-C 1g/m2 q12h days 1-3, idarubicin 10mg/m2 days 2-3;
  3. and 3 quarterly reinduction courses during maintenance including Ara-C 80mg/m2 days 1-5, CCNU 40mg and mitoguazone 350mg/m2 day 1, ± fludarabine days 1-2.
  Interventions: Drug: Active comparator (no fludarabine)
- 2 (Experimental): Fludarabine arm
  The same regimen with fludarabine 20 mg/m2/day IV for 30 minutes
  1. induction course + fludarabine days 2-7;
  2. consolidation course + fludarabine days 4-5;
  3. during reinduction courses + fludarabine days 1-2.
  Interventions: Drug: Experimental (fludarabine)

INTERVENTIONS:
Drug: Active comparator (no fludarabine) — 1. Ara-C (100 mg/m2/d by continuous IV infusion 7 days), idarubicin (8 mg/m2/d (IV) for 5 days), GM-CSF a dose of 5 mg/kg/d on day 1. (Novartis Laboratory, Rueil-Malmaison, France).
  2. The consolidation course: intermediate-dose Ara-C (1g/m2 g 3-hour infusion twice a day 1 through 3) and idarubicin (10 mg/m2 on days 4 through 5). In the allocated arm
  3. Maintenance therapy for one year with 6-thioguanine (100 mg/m2/d orally on days 1 through 4 every week, Ara-C (60 mg/m2 SC on day 5 weekly) interrupted every 3 months with a reinduction course including CCNU (40 mg orally on day 1), mitoguazone (350 mg/m2 on day 1) and Ara-C (40 mg/m2 sc twice daily day 1 to 5)
  Other Names: Arm A
  Arms: 1
Drug: Experimental (fludarabine) — The same regimen with addition of fludarabine in every treatment sequence
  1. Induction course: Fludarabine (20 mg/m2/d, IV for 30 minutes) was started in the assigned group on day 2 and continued until the end of cytarabine treatment on day 7.
  2. Consolidation course: In the allocated arm, fludarabine (20 mg/m2/d, IV) was administered on days 2 through 3, 4 hours prior to cytarabine infusion.
  3. Reinduction courses: Ara-C associated in the allocated group with fludarabine (20 mg/m2/d, IV) on days 1 through 2.
  Other Names: Arm B
  Arms: 2

SUMMARY:
In this study, patients were randomly assigned to either receive fludarabine or not (20 mg/m2/d) in addition to induction chemotherapy, consolidation chemotherapy and the 3 subsequent re-induction courses during maintenance.

DETAILED DESCRIPTION:
Eligibility for enrollment in the study was limited to patients aged 60 to 75 years old with previously untreated de novo AML as defined morphologically by the French-American-British (FAB) classification with the exception of M3 and M7 subtypes.10,11 The bone marrow aspirate had to show at least 30 percent of nonerythroid blast cells. Patients were not eligible if they had a performance status before diagnosis of 2 or more according to the World Health Organization (WHO) grading system, congestive heart failure or abnormal left ventricular ejection fraction, severe hepatic or renal disturbances if not related to leukemia (hepatic enzymes levels over four times the normal values, serum bilirubin over 35 micromol/L, creatinine over 150 micromol/L). Patients with previous unexplained cytopenia were eligible for the study. Conversely, patients with a history of documented myelodysplastic or myeloproliferative syndrome or previously treated with chemotherapy or radiation could not enter the study. The study received in June 1996 approval from the ethics' board of the Nancy Hospital and written informed consent was given by all eligible patients before entering the study, in accordance with the Declaration of Helsinki. The enrollment period was open from November 1996 to April 2000.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 60 to 75 years old
* untreated de novo AML
* performance status less than 2

Exclusion Criteria:

* performance status more than 2
* congestive heart failure or abnormal left ventricular ejection fraction
* severe hepatic or renal disturbances
* history of documented myelodysplastic or myeloproliferative syndrome
* patients previously treated with chemotherapy or radiation

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 1996-06; Primary Completion 2000-04 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Event-free survival (EFS) | long term results (median follow up: 71 months)

SECONDARY OUTCOMES:
evaluation of the CR rate, remission duration disease-free survival (DFS) overall survival (OS), | long term results (median follow up: 71 months)

CONTACTS AND LOCATIONS:
Overall Officials: Francis WITZ, MD, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- GOELAMS, Tours, France